CLINICAL TRIAL: NCT06639659
Title: Bilateral Supra-Zygomatic Sphenopalatine Ganglion Block Versus Dexmedetomidine for Relief of Postoperative Pain and Surgical Field Improvement in Trans-nasal Endoscopic Pituitary Surgery
Brief Title: Sphenopalatine Block vs Dexmedetomidine Infusion in Trans Nasal Endoscopic Pituitary Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: sphenopalatine block in TEPS
Record Dates: First submitted 2024-09-26; First posted 2024-10-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-09

CONDITIONS: Sphenopalatine Ganglion Nerve Block; Transnasal Endoscopic Pitutary Surgery
MeSH Terms: interventions — Sphenopalatine Ganglion Block; Dexmedetomidine; Anesthesia, General; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (control group) (n=23) patients will be operated under general anesthesia. (Placebo Comparator)
  Interventions: Other: General Anesthesia (control group)
- Group SPGP (n=23) patients will receive ultrasound guided bilateral sphenopalatine block (Active Comparator)
  Interventions: Procedure: Sphenopalatine Ganglion Block
- Group DEX (n=23) patients will receive dexmedetomidine drug. (Active Comparator)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion Block — patients will receive ultrasound guided bilateral supra-zygomatic sphenopalatine ganglion block.
  Arms: Group SPGP (n=23) patients will receive ultrasound guided bilateral sphenopalatine block
Drug: Dexmedetomidine — patients will receive 1 µg/kg dexmedetomidine within 10 minutes, followed by maintenance dose throughout the surgery.
  Arms: Group DEX (n=23) patients will receive dexmedetomidine drug.
Other: General Anesthesia (control group) — patients will be operated under general anesthesia including routine protocol for these cases
  Arms: Group C (control group) (n=23) patients will be operated under general anesthesia.

SUMMARY:
Improving pain and surgical field by using sphenopalatine ganglion block and dexmedetomidine in trans-nasal endoscopic pituitary surgery.

DETAILED DESCRIPTION:
Pituitary neoplasm is one of the most common sellar pathology. Trans-nasal endoscopic pituitary surgery (TEPS) evolved rapidly, almost replacing the craniotomy approach. TEPS, a surgical instrument, is primarily executed through a minimally invasive approach through the nostril to access a pituitary tumor.

That is why the anesthetic plan must ensure the best possible surgical field visualization and the most adequate analgesia.

Multimodal anesthesia including regional and general anesthesia are obtained to optimize surgical field by decreasing bleeding, reduce pain, promote rapid recovery and potential economic gains for the hospital.

The sphenopalatine ganglion block (SPGB) is considered one of the regional anesthetic techniques that is safe and easy anesthetic procedure used to control bleeding and for postoperative analgesia.

Dexmedetomidine (DEX) has become popular for induced hypotension. It is an α2-adrenoceptor agonist with a sympatholytic and analgesic effect. It provides a unique conscious sedation without respiratory depression. It is used effectively in optimizing surgical field through its hemodynamic stability effect.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 21-64 years old.
* sex: males and females.
* Body mass index: 35 kg/m2.
* ASA Physical status: grade Ⅰ-Ⅱ.

Exclusion Criteria:

* patients receiving beta blockers, anti-coagulants and antihypertensive medications also patients receiving clonidine or benzodiazepines, neuroleptics or antidepressants two weeks prior to the study.
* Any contraindication for regional anesthesia e.g. coagulopathy, infection at site of block and hypersensitivity to any drug used in this study.
* Patients who are known to be drug addict.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain using VAS scale. | 24hours
  Pain will be assessed based on VAS scale from (1-10), as 1 is the least pain and 10 is the maximal pain possible at 2, 4, 6, 12 and 24h after surgery.
Surgical field using Average Category Scale (ACS). | 5hours
  Done by asking the surgeon about amount of bleeding on a scale of (0-5) as 0= no bleeding and 5= sever bleeding, every 15 min interval till the end of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig Univesity Hospital, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Anthony Cometa M, Zasimovich Y, Smith CR. Percutaneous sphenopalatine ganglion block: an alternative to the transnasal approach. Int J Obstet Anesth. 2021 Feb;45:163-164. doi: 10.1016/j.ijoa.2020.10.002. Epub 2020 Oct 17. No abstract available. PMID 33199256
- [Result] Mantovani G, Sgarbanti L, Indaimo A, Cavallo MA, De Bonis P, Flacco ME, Scerrati A. Effects of a sphenopalatine ganglion block on postcraniotomy pain management: a randomized, double-blind, clinical trial. Neurosurg Focus. 2023 Dec;55(6):E13. doi: 10.3171/2023.9.FOCUS23549. PMID 38262005
- [Result] Hutton M, Brull R, Macfarlane AJR. Regional anaesthesia and outcomes. BJA Educ. 2018 Feb;18(2):52-56. doi: 10.1016/j.bjae.2017.10.002. Epub 2017 Nov 27. No abstract available. PMID 33456810